CLINICAL TRIAL: NCT07060157
Title: Comparative Efficacy of Resveratrol 1 % Gel and Trichloroacetic Acid 20% in Treatment of Melasma: A Split-face Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amira Mohamed Bakry Refaay, doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: resveratrol in melasma
Record Dates: First submitted 2025-03-21; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Melasma
Keywords: resveratrol in melasma
MeSH Terms: conditions — Melanosis | interventions — Resveratrol; Gels

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Active Comparator): left side of face the patient will be given resveratrol 1 % gel once daily at night (homThee use ).
  Interventions: Drug: resveratrol 1 % gel
- Group B (Active Comparator): The right side of face will treated with TCA20% every two weeks for 3months.
  Interventions: Drug: TCA20%

INTERVENTIONS:
Drug: resveratrol 1 % gel — left side of face the patient will be given resveratrol 1 % gel once daily at night (Home use ).
  Other Names: 1
  Arms: Group A
Drug: TCA20% — left side of face the patient will be given resveratrol 1 % gel once daily at night (homThee use ).
  Arms: Group B

SUMMARY:
1. To evaluate the efficacy and safety of topical resveratrol 1 % gel in treatment of melasma.
2. To compare between the efficacy of topical resveratrol 1 %gel versrs chemical peeling with TCA 20% in melasma.

DETAILED DESCRIPTION:
Melasma is a chronic, acquired disorder of focal hypermelanosis. It clinically presents as hyperpigmented patches over photo-exposed areas (Espósito.,et al 2022). Melasma classified clinically into; Centrofacial, malar, mandibular, indeterminate , and extrafacial types . By wood's lamp ,melasma classified into epidermal, dermal, and mixed forms (Putra Gofur N et al . , 2021) .

Chronic ultraviolet (UV) exposure, genetic factors, and sex hormones are generally believed to be involved in the occurrence of melasma. Other factors implicated are phototoxic drugs, anticonvulsant medications, and the use of certain cosmetics (Ortonne et al., 2009).

Treating melasma is challenging especially in patients with dark skin types , classified as Fitzpatrick types IV to VI, due to the possibility of relapse and susceptibility to post-inflammatory hyperpigmentation (PIH) (Rodrigues and Pandya., 2015).

Although various therapeutic approaches including pharmacological and procedural treatments have been considered in melasma management, none of them is completely satisfactory (Rodrigues and Pandya., 2015).

Ongoing clinical trials continue to explore new topical treatment options for melasma, aiming to develop more effective and safer alternatives with fewer side effects. Traditional agents like hydroquinone remain the gold standard, but concerns over irritation and potential long-term risks have driven research into novel formulations. (Christian and Michelle.,2024) .

Resveratrol is a natural phenolic compound present in wide variety of foods, such as grapes, blueberries and peanuts . It has shown many bioactivities, such as antioxidant, anti-inflammatory, immunomodulatory and anticancer agent (Athar M., 2009).

Resveratrol a direct tyrosinase inhibitor by it is ability to bind to the active site of tyrosinase and interfere with its ability to catalyze the conversion of tyrosine to melanin. This could be achieved by interacting with the copper ions present at the enzyme's active site, which are critical for its enzymatic function. Resveratrol has also an indirect inhibitor by modulation the expression of genes involved in melanin synthesis. It has been shown to affect various signaling pathways, including those related to the melanogenesis process, such as the MITF (microphthalmia-associated transcription factor) pathway. By downregulating these pathways, resveratrol can reduce the production of tyrosinase, thus decreasing melanin synthesis. Furthermore, it can affect keratinocytes, which regulate the function of melanocyte (Newton et al., 2007).

Resveratrol regulates the inflammatory process of keratinocytes and protects them from oxidative damage. In this way, it prevents keratinocyte-induced melanocyte stimulation. Furthermore, it has a rescuing effect on the stemness of interfollicular epidermal cells that can repair signs of photoaging in the melasma (Na J et al., 2019).

Chmical peels are an attractive treatment option for patients, as they are an affordable in-office procedure, quick in achieving results, and the patient can return to daily activities immediately after the procedure (Rendon et al., 2010).

Chemical peels are typically categorized based on their depth of skin penetration, which can range from light to medium to deep. Several factors, including pH and concentration, application technique, and the patient's skin condition and sensitivity, influence the extent of the therapeutic effects (O'Connor A A .,et al 2018).

Trichloroacetic Acid (TCA) is a versatile peeling agent, since the peel depth can be varied according to the concentration of TCA solution used. It is commonly used as a superficial to medium depth peel with advantages of being stable, inexpensive, self-neutralizing and without any systemic toxicity (Rubin MG et al., 2018)

ELIGIBILITY:
Inclusion Criteria:

* • Age: 18-50 years old.

  * Pattern of melasma: Bilateral symmetrical facial melasma of any pattern.
  * Fitzpatrick skin phototypes: Types III, IV and V.

Exclusion Criteria:

* Pregnancy and lactation.

  * Patients taking oral contraceptive pills, hormonal replacement therapy or treatment for chronic illness at the time of the study or during the past 6 months.
  * Coexistence of diseases associated with hyperpigmentation such as Addison disease.
  * History of Scarring and keloid tendency
  * Active skin infections as active HSV.
  * Previous history of post- inflammatory hyperpigmentation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 41 (Estimated)
Dates: Start 2025-07-22 (Estimated); Primary Completion 2026-08-08 (Estimated); Study Completion 2027-06-08 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is the change in hemi-Melasma Area and Severity Index (hemi-MASI) score from baseline to one month after the end of treatment (follow-up) | 3 months
  assessed by clinical evaluation and photographic documentation. Clinical efficacy will be categorized as:
  Excellent response: >75% decrease in hemi-MASI score
  Very good response: 50-75% decrease in hemi-MASI score
  Good response: 25-50% decrease in hemi-MASI score
  Poor response: <25% decrease in hemi-MASI score

CONTACTS AND LOCATIONS:
Locations (1):
- Assuit, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes